CLINICAL TRIAL: NCT06630598
Title: The Effects of the ©Violence, Evidence, Guidance, and Action (VEGA) Family Violence Education Resources on Canadian Clinical Psychology Students' Attitudes, Knowledge, and Behaviours
Brief Title: Impacts of the VEGA Family Violence Education Resources for Psychology Trainees
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Elisa Romano, Professor, University of Ottawa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: H-06-24-10490
Record Dates: First submitted 2024-09-30; First posted 2024-10-08 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Family Violence
Keywords: Intimate Partner Violence; Child Maltreatment; Family Violence; Health Professions Education

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to a training group or a wait-list control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- VEGA Family Violence Education Resources (Experimental): Students in this arm will receive access to the online VEGA Family Violence Education Resources and will be asked to complete modules covering information about family violence in Canada, creating safety for survivors in clinical settings, recognizing and responding to child maltreatment and intimate partner violence, three interactive learning scenarios, and voices of those with lived experiences of family violence.
  Interventions: Behavioral: Online Family Violence Education Resource
- No Training (No Intervention): Students in this arm will not receive access to the training until the end of the pre- and post-training data collection for the Arm 1 group.

INTERVENTIONS:
Behavioral: Online Family Violence Education Resource — The VEGA Family Violence Education Resources (© 2020 VEGA Project, McMaster University) is an on-line suite of educational resources that target professionals who are likely to encounter survivors of family violence in professional and clinical settings. The resources provide information about family violence, appropriate clinical responses, legal obligations, and more. The resources are broken down into several training modules and include three interactive learning scenarios. The training modules include:
  Know About Family Violence in Canada Creating Safety Recognizing and Responding Safely to Child Maltreatment Recognizing and Responding Safely to Intimate Partner Violence Voices of those with Lived Experiences of Family Violence
  Arms: VEGA Family Violence Education Resources

SUMMARY:
The current research project aims to assess the effectiveness of the ©Violence, Evidence, Guidance, and Action (VEGA) Family Violence Education Resources (VEGA Project, 2019) in improving the knowledge, self-efficacy, and clinical responses of clinical psychology doctoral students to family violence in clinical settings. The VEGA on-line training is a collection of family violence online education resources designed to inform health and social service practitioners about family violence in a Canadian context, including definitions of family violence, mandatory reporting duties, effective responding to survivors, and more. Participants in this trial will be doctoral students recruited from accredited Clinical Psychology programs across Canada. Participants will be assigned to an intervention or wait-list control group, and the outcome measures consist of knowledge and attitudes about family violence, as well as measures of skills relevant to appropriately responding to survivors in clinical settings. Further, participants will be invited to complete a qualitative interview after the intervention to discuss overall impressions of the training and other ways the training changed their perspectives, if at all, on family violence.

DETAILED DESCRIPTION:
The goal of the current research is to conduct a randomized controlled trial of the ©Violence, Evidence, Guidance, and Action (VEGA), Family Violence Education Resources (VEGA Project, 2019) among a sample of clinical psychology graduate students across Canadian universities to assess whether it is effective in improving responses to child maltreatment and intimate partner violence (IPV) (collectively referred too throughout as "family violence") in clinical settings. For this study, students belonging to accredited Clinical Psychology doctoral programs from Canadian universities will be randomized into either (a) an intervention group that will complete the online VEGA Family Violence Education Resources, OR (b) a control group who will not complete the training (but who will have the opportunity to do so following the completion of outcome data collection ; wait-list control). Throughout this evaluation study, a variety of pre- and post-training outcome measures will be administered participants; these measures are intended to assess reactions to the training, changes in family violence knowledge, changes in attitudes toward IPV and child maltreatment, and clinically relevant behaviours in responding to suspicions and disclosures of family violence by clients/patients in clinical practice settings. After completing the measures and the training, a subset of randomly selected students from the intervention group will be invited to participate in a one-on-one qualitative interview with a member of the research team via Zoom, during which they will be asked to share their perspectives on the training and how it impacted/may impact their work (or not) with clients who have experienced IPV and/or child maltreatment. Information provided from the quantitative measures and qualitative interviews will allow us to answer the following questions: (1) Was the training engaging and relevant to clinical psychology students? (2) Was the training able to improve the knowledge and self-efficacy of students regarding family violence? (3) Was the training able to change behaviours and improve the response of clinical psychology students to clients (or future clients) experiencing family violence in their professional training settings? Note: Used with permission from © 2020 VEGA Project, McMaster University. All rights reserved. All questions regarding the use and evaluation of the VEGA Family Violence Education Resources, or the VEGA Project more generally, should be directed to Dr. Melissa Kimber at vega@mcmaster.ca

ELIGIBILITY:
Inclusion Criteria:

* Be a student in the Clinical Psychology graduate program of a Canadian university.
* Be engaged in clinical work as part of program requirements
* Speak and read English
* Have internet access

Exclusion Criteria:

-Currently participating in any other training relating to child maltreatment or intimate partner violence outside of mandatory or elective course material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-10-30 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Changes in perceived knowledge and preparedness, and opinions about family violence as measured by the Modified Provider Readiness to Manage Intimate Partner Violence Survey Items (Modified PREMIS) | Week one (pre-training), and again Week four (post-training)
  Changes in self-rated Knowledge/Preparation and Opinions about intimate partner violence and child maltreatment. Perceived preparedness to manage intimate partner violence and child maltreatment (14 items, 7-point Likert scale ranging from &amp;#34;Not Prepared&amp;#34; to &amp;#34;Quite Well Prepared&amp;#34;). Perceived Knowledge about intimate partner violence and child maltreatment (22 items, 7-point Likert scale ranging from &amp;#34;Nothing&amp;#34; to &amp;#34;Very Much&amp;#34;). Opinions about intimate partner violence and child maltreatment (47 items, 4-point Likert scale, ranging from &amp;#34;Strongly Agree&amp;#34; to &amp;#34;Strongly Disagree&amp;#34;).
Reactions - Interest and Relevancy of Intervention Material | During Weeks two through three - completed during training period
  Measurement of participant reactions to training contents, specifically in terms of the learning objectives and relevancy of each individual training module in order to examine engagement and interest. Agreement on whether training modules met their learning objectives, and whether training module content was relevant is measured on a 7-point scale from Strongly Agree to Strongly Disagree.
Changes in VEGA content knowledge | Week one (pre-training), and again Week four (post-training)
  Changes in knowledge regarding family violence content in VEGA modules. Content knowledge measure contains 34 multiple choice questions about the VEGA Family Violence Education Resources. Each question has a maximum score of 1, and minimum score of 0, for a total range of 0 to 34.
Performing relevant clinical behaviours in clinical settings with clients, as measured by a Behavioural Checklist | One month post-training.
  A checklist of a variety of clinically-relevant behaviours that are recommended and suggested as best practice when working with a survivors of family violence. Participants indicate whether or not they have engaged in certain behaviours. Participants may also indicate if they have not had the opportunity to engage in selected behaviours. The checklist covers 72 clinical actions relating to the VEGA family violence resources, with participants being able to select &#34;Yes&#34;, &#34;No&#34;, or &#34;N/A&#34; for each action performed in the previous 30 days.

SECONDARY OUTCOMES:
Changes in attitudes towards evidence-based practice and interventions as measured by the Evidence-Based Practice Attitude Scale (EBPAS) | Week one (pre-training), and again Week four (post-training)
  Changes ttitudes toward utilizing evidence-based interventions and their importance in professional and clinical settings. Measured with the EBPAS (Evidence-Based Practice Attitude Scale) - fifteen items across four subscales (Requirements, Appeal, Openness, and Divergence) measured on four-point Likert scales ("Not at All" to "To a Very Great Extent").
Interview on experiences with the VEGA family resources | One month post-training.
  A randomly selected subset of participants will be invited to participate in an interview one month after the training to discuss their opinions on the VEGA Family Violence Education Resources, what they learned (if anything), and how their clinical approaches have changed.

CONTACTS AND LOCATIONS:
Overall Officials: Elisa Romano, PhD, Clinical Psychology, Principal Investigator — University of Ottawa
Locations (1):
- University of Ottawa - Child Wellbeing Lab, Ottawa, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No